CLINICAL TRIAL: NCT02335151
Title: Resectable Pancreatic Adenocarcinoma - Does the Type of Anesthesia Have an Impact on Circulating Tumor Cells?
Brief Title: CTC Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Winterthur KSW (Other); Triemli Hospital (Other); Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016 -00448
Record Dates: First submitted 2014-12-13; First posted 2015-01-09 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Adenocarcinoma; Circulating Tumor Cells; Pancreatic Neoplasms
Keywords: Circulating Tumor Cells; Anesthesia and immunity; Cell Search System
MeSH Terms: conditions — Adenocarcinoma; Neoplastic Cells, Circulating; Pancreatic Neoplasms | interventions — Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane (Experimental): General anesthesia with Desflurane
  Interventions: Drug: Desflurane
- Propofol (No Intervention): General anesthesia with Propofol

INTERVENTIONS:
Drug: Desflurane — Apply desflurane as anesthetic
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
Proportion of circulating tumor cells (CTC) in the postoperative phase after curative tumor removal of pancreatic cancer will be determined and correlated to the accordance of anesthesia (desflurane versus propofol)

DETAILED DESCRIPTION:
This prospective, randomized study will be conducted over a 36-month period to investigate whether commonly used anesthetics (volatile versus intravenous) have an effect on the changes or occurrence of CTC in patients suffering from primary pancreatic cancer undergoing curative surgery. The specific research question is if there are changes of the CTC count in the postoperative phase in the desflurane group (intervention) compared to the propofol one (control). A secondary question is if these changes can be correlated to tumor outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85
* ASA I-III ( American Society of Anesthesiologists)
* Resectable pancreatic adenocarcinoma
* Primary surgery
* No neoadjuvant therapy
* Written informed consent

Exclusion Criteria:

* Metastatic disease
* Other than primary surgery (recurrence, reconstruction)
* Pre-operative chemotherapy
* Chronic opioid use
* Known hypersensitivity or suspected allergy to propofol, soya or egg proteins
* Known hypersensitivity to volatile anaesthetics (malignant hyperthermia)
* Pregnancy
* Breast feeding
* Enrolment in any other clinical trial during the course of this trial, 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Peak of CTC in the postoperative phase after curative tumor removal | Day 0 to Day 7
  CTC will be counted and peak of CTC will be determined.

SECONDARY OUTCOMES:
Kinetics of CTC after surgery up to day 7 | 1 year
  CTC will be counted and kinetics of CTC will be determined.
Month to Tumor recurrence | 1 year
  Tumor recurrence will be monitored.
Number of surviving patients | 1 year
  One year after surgery the number of patients still being alive will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof. MD, Principal Investigator — University of Zurich
Locations (4):
- Switzerland (4):
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No
Data will not be shared